CLINICAL TRIAL: NCT01998230
Title: Early Oral Feeding Following Thoracolaparoscopic Oesophagectomy in Patients With Esophageal Cancer: a Randomized Clinical Trial
Brief Title: Early Oral Feeding Following Thoracolaparoscopic Oesophagectomy in Patients With Esophageal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yin Li (Other Government)
Responsible Party: Sponsor-Investigator, Yin Li, Vice President of Henan Cancer Hospital, Henan Cancer Hospital
Organization: Henan Cancer Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH
Record Dates: First submitted 2013-11-15; First posted 2013-11-28 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; esophagectomy; oral feeding
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early oral feeding group (Experimental): In this goup patients with esophagectomy are encouraged to begin the oral intake carefully and adjust according to tolerance on post operative day 1.
  Interventions: Dietary Supplement: early oral feeding
- Delayed oral feeding group (No Intervention): In delayed oral feeding group the patients receive isotonic saline by the nasoenteral feeding tube at 20 mL/h until the morning of post operative day1. Nutrition was then commenced at 20 mL/h. The rate was increased by 20 mL/h each day if tolerated, up to 80 mL/h.Esophagography was performed on postoperative day 7. Sip of water were allowed after confirming the absence of anastomosis leakage, and a full liquid diet was implemented on the following day and enteral infusion halted.

INTERVENTIONS:
Dietary Supplement: early oral feeding — In the early oral feeding group, the patients are encouraged to intake liquid food on post operative day 1.
  Arms: Early oral feeding group

SUMMARY:
The purpose of this study is to determine the feasibility of early oral food intake postoperatively in patients with thoracolaparoscopic esophagectomy. More and more evidence confirmed the role of early early enteral nutrition (NE) after esophagectomy in patients with esophageal cancer. Although enteral catheter feeding has been shown to be beneficial in patients with esophagectomy, the preference for this modality also rests on the traditional but undocumented reluctance to allow food at will. These assumed hazards of allowing normal food in the immediate postoperative period have not been scientifically tested and should be viewed against both the benefits and side effects of any artificial feeding modality. Whether early oral feeding after esophagectomy affects the incidence of life-threatening surgical complications, shortens the recovery time of bowel function and the postoperative hospital stay, improves postoperative quality of life in comparison with artificial feeding modality remains unclear. The investigators compared a routine of allowing liquid food at will from the first day after surgery with a routine of nil-by-mouth and enteral nutrition for the first 7 postoperative days. The main endpoint is the incidence rate of complications.

DETAILED DESCRIPTION:
The literature concludes that patients should be allowed food without delay (at will) after colorectal surgery and that the customary withholding of oral intake (nil-by-mouth) for the first postoperative days is unnecessary. Robust data also suggest that the investigators should avoid the nil-by-mouth regimen after major gynecologic, urologic, and vascular surgery. The safety of early oral feeding after esophagectomy has not been investigated previously.In 2008, the results of a randomized multicenter clinical trial investigating whether a routine of allowing normal food at will immediately increases morbidity after major upper gastrointestinal surgery showed that allowing patients to eat normal food at will from the first day after major upper gastrointestinal surgery does not increase morbidity compared with traditional care with nil-by-mouth and enteral feeding. The assumed hazards of allowing oral food intake in the immediate postoperative period in patients with esophagectomy have not been scientifically tested and should be viewed against both the benefits and side effects of any artificial feeding modality.

This is a randomized study investigating the role of early oral feeding in patients with esophagectomy.In the early oral feeding group nasogastric tube is not placed routinely and patients are encouraged to intake liquid food on postoperative day 1 (POD1). In delayed oral feeding group the patients receive isotonic saline by the nasoenteral feeding tube at 20 mL/h until the morning of POD 1. Nutrition was then commenced at 20 mL/h. The rate was increased by 20 mL/h each day if tolerated, up to 80 mL/h. Esophagography is performed on postoperative day 7. Sip of water were allowed after confirming the absence of anastomotic leakage, and a full liquid diet was implemented on the following day and enteral infusion halted. The complications defined in previous study and bowel function and recovery were recorded carefully. The primary end point of this study is the postoperative complications and the secondary end points are quality of life,bowel function recovery time and length of postoperative stay between the two groups. The investigators estimated the minimum rate of patients with complications in control group population at 23%. An increase of this to 36% was considered clinically important. Detecting a difference of this magnitude or greater at a level of statistical significance of 0.05 and a power of 0.90 with a one-tailed test of proportions required a total of 130 patients in each group.Considering the rate of drop-out a total of 280 patients will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

Adults subject to thoracolaparoscopic esophagectomy for esophageal cancer.

Exclusion Criteria:

Stage investigations indicating unresectable advanced disease(T4 or M1a,M1b). Patients with any other serious underlying medical condition that would impair the ability of the patient to receive or comply with protocol treatment.

Patients with unstable situation after surgery (eg, need ventilation and ICU treatment) Patients medically unfit for surgical resection. Patients with pulmonary reserve inadequate to undergo thoracotomy and extensive mediastinal lymphadenectomy.

Mentally disabled. Expected life duration of less than 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Postoperative complication | an expected average of 4 weeks
  postoperative complications are graded according to Clavin-Dindo grading system

SECONDARY OUTCOMES:
Quality of Life assessment | 6 months
Length of postoperative stay | an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yin Li, Principal Investigator — Henan Cancer Hospital (The Affiliated Cancer Hospital of Zhengzhou University)
Locations (1):
- Henan Cancer Hospital (The Affiliated Cancer Hospital of Zhengzhou University), Zhengzhou, Henan, China

REFERENCES:
- [Derived] Chen X, Wang P, Leng C, Sun H, Liu X, Zhang R, Qin J, Hua X, Yu Y, Li H, Zhang J, Wu Z, Li Y. Early oral feeding after esophagectomy accelerated gut function recovery by regulating brain-gut peptide secretion. Surgery. 2022 Sep;172(3):919-925. doi: 10.1016/j.surg.2022.04.041. Epub 2022 Jul 3. PMID 35794044
- [Derived] Yang F, Li L, Mi Y, Zou L, Chu X, Sun A, Sun H, Liu X, Xu X. Effectiveness of the Tailored, Early Comprehensive Rehabilitation Program (t-ECRP) based on ERAS in improving the physical function recovery for patients following minimally invasive esophagectomy: a prospective randomized controlled trial. Support Care Cancer. 2022 Jun;30(6):5027-5036. doi: 10.1007/s00520-022-06924-8. Epub 2022 Feb 22. PMID 35190895
- [Derived] Sun HB, Li Y, Liu XB, Wang ZF, Zhang RX, Lerut T, Zheng Y, Liu SL, Chen XK. Impact of an Early Oral Feeding Protocol on Inflammatory Cytokine Changes After Esophagectomy. Ann Thorac Surg. 2019 Mar;107(3):912-920. doi: 10.1016/j.athoracsur.2018.09.048. Epub 2018 Nov 4. PMID 30403976